CLINICAL TRIAL: NCT05232045
Title: Automated System for Monitoring Urine Output in Intensive Care Patients: What Are the Advantages? Before-after Intervention Study
Brief Title: Automated System for Monitoring Urine Output in Intensive Care Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0033-22-MMC
Record Dates: First submitted 2022-02-01; First posted 2022-02-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury in the ICU

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Automated urinary output collection system group (tight monitoring of urine output)
  Interventions: Drug: Automated urinary output collection system group (tight monitoring of urine output)
- Manual urinary output collection system group (routine monitoring of urine output)

INTERVENTIONS:
Drug: Automated urinary output collection system group (tight monitoring of urine output) — Automated urinary output collection system group (tight monitoring of urine output)
  Groups: Automated urinary output collection system group (tight monitoring of urine output)

SUMMARY:
Acute kidney injury is common among ICU-admitted patients, and is associated with increased morbidity and mortality. Early recognition is essential to prevent complications. In this study we aim to examine whether strict monitoring of urine output may reduce the incidence of acute kidney injury, allow for less positive fluid balance and reduce the clinical symptoms of fluid overload in ICU patients. Currently we monitor urine output using a Urinometer, with manual recording. From June 2022 we will begin routine use of an automated urine monitoring system in the ICU and test its effect on the parameters listed above. We will conduct a before-after retrospective intervention. The group of patients in whom the automated system will be used, from June 2022 to January 2024, will be the study group. The patients admitted to the ICU in the period between January 2021 and June 2022 will be the control group. We will include patients aged 18-100, who were admitted to the General Intensive Care Unit in Meir Medical Center from January 2021 to January 2024, and had admission time longer than 48 hours. Patients without a urinary catheter will not be included. The study will be conducted in the format of observational data collection from hospital files and computerized systems (Metavision system and Chameleon system). We estimate that we will include about 900 patients in the study group and about 900 in the control group. All demographic and inpatient data will be statistically examined by a qualified statistician depending on the type of data.

ELIGIBILITY:
Inclusion Criteria: Patients aged 18-100, who were admitted to the General Intensive Care Unit in Meir Medical Center from January 2021 to January 2024, and had admission times longer than 48 hours.

-

Exclusion Criteria: Patients without a urinary catheter, Patients with admission times less than 48 hours.

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-100, who were admitted to the General Intensive Care Unit in Meir Medical Center from January 2021 to January 2024
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of acute kidney injury | June 2023-January 2024
  Primary outcome: To investigate whether the use of an automatic urinary output monitoring system in ICU patients will decrease the incidence of acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No